CLINICAL TRIAL: NCT01462162
Title: A Prospective Observational Study to Evaluate and Correlate the Impact of Treatment With Tocilizumab (RoActemra®) on Fatigue and Different Factors Influencing Fatigue in Participants With Rheumatoid Arthritis in Routine Clinical Practice
Brief Title: A Prospective Observational Study of Tocilizumab (RoActemra/Actemra) in Participants With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27833
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA) who have been considered and proposed by the rheumatologist to start treatment with Tocilizumab (RoActemra) according to the indications of the summary of product characteristics of the product and the standard clinical practice of each participating center will be followed-up for 6 months.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: RoActemra; Actemra

SUMMARY:
This prospective observational study will investigate the effect of tocilizumab on fatigue in participants with moderate to severe rheumatoid arthritis who have an inadequate response to disease-modifying antirheumatic drugs or anti-tumour necrosis factor (anti-TNF) drugs. Data will be collected from participants for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe RA who have been considered and proposed by the rheumatologist to start treatment with Tocilizumab according to his/her clinical judgment and the conditions approved in the Summary of Product Characteristics (SPC).

Exclusion Criteria:

* Participants previously or currently treated with RoActemra/Actemra in clinical trials
* Absolute neutrophil count less than or equal to (</=) 2x10^9 per liter (/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Spain (14):
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Mollet del Vallès, Barcelona
  - Sabadell, Barcelona
  - Sant Joan Despí, Barcelona
  - Girona, Girona
  - A Coruña, La Coruña
  - Lugo, Lugo
  - Cartagena, Murcia
  - El Palmar, Murcia
  - Lorca, Murcia
  - Ourense, Orense
  - Vigo, Pontevedra
  - Tarragona, Tarragona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 122 participants were recruited, 2 participants were excluded from analysis, one due to non-compliance with the inclusion criteria and other due to compliance with the exclusion criteria.
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA) who had been considered and proposed by rheumatologist to start treatment with tocilizumab (RoActemra) according to the indications of the summary of product characteristics and the standard clinical practice of each participating center were followed-up for 6 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Participants
Started | 120
Completed | 108
Not Completed | 12
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 4
Not completed — Abnormal laboratory parameters | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All participants who satisfied inclusion and exclusion criteria of the study were included in the analysis.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Regression Coefficient Between Change in Fatigue Score as Measured by the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) at Week 12 and Change in Main Variables at Week 12
Description: Regression analysis between change in FACIT-F scale and change in following variable were assessed: DAS28-ESR (total score range: 0-9.4, higher score=more disease activity), Epworth sleepiness scale (total score range: 0-24, higher score=higher degree of sleepiness), back depression inventory (total score range: 0-63, score higher than 18 indicates moderate to severe symptoms of depression). The total score of the FACIT-F questionnaire ranges from 0=worse score to 52=better score. Regression coefficient (R) and coefficient of determination (R^2) were calculated. Difference (1-R^2)=the variation in the changes in fatigue not explained by independent variables, that is, independent contribution of these changes in fatigue to the assessment of RA. Only variables with available data were reported.
Time Frame: Week 12
Population: Effectiveness analysis population included all participants who had all measurements of effectiveness and had complete information of the FACIT questionnaire throughout the study. Here, Number of participants analyzed (N) = number of participants evaluable for this measure.
Measure: Number; unit: unstandardized regression coefficient
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 65
unstandardized regression coefficient
  DAS-28 | -2.200
  Sleepiness | -0.944
  Depression | -0.707
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in DAS-28 score; Test type: Superiority or Other; p = 0.006, Regression, Linear
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in sleepiness score; Test type: Superiority or Other; p = 0.000, Regression, Linear
Statistical Analysis 3: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in depression score; Test type: Superiority or Other; p = 0.000, Regression, Linear

2. Primary Outcome: Regression Coefficient Between Change in Fatigue Score as Measured by the FACIT-F at Week 24 and Change in Main Variables at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Effectiveness analysis population. Here, N=number of participants evaluable for this measure.
Measure: Number; unit: unstandardized regression coefficient
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA) who have been considered and proposed by the rheumatologist to start treatment with Tocilizumab (RoActemra) according to the indications of the summary of product characteristics of the product and the standard clinical practice of each participating center were followed-up for 6 months.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 71
unstandardized regression coefficient
  DAS-28 | -1.743
  Sleepiness | -0.990
  Depression | -0.658
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in DAS-28 score; Test type: Superiority or Other; p = 0.023, Regression, Linear
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in sleepiness score; Test type: Superiority or Other; p = 0.007, Regression, Linear
Statistical Analysis 3: Comparison: Rheumatoid Arthritis Participants; change in fatigue score versus change in depression score; Test type: Superiority or Other; p = 0.000, Regression, Linear

3. Secondary Outcome: Change From Baseline to Week 12 and 24 in Fatigue Score as Assessed by FACIT-F
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline, Week 12, Week 24
Population: Effectiveness analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 85
units on a scale
  Baseline | 26.8 (12.4)
  Change at Week 12 | 4.6 (10.4)
  Change at Week 24 | 5.4 (11.2)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Change From Baseline to Week 12 and 24 in Serum Hemoglobin
Description: The hemoglobin level was measured in grams per liter (g/L). Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure. n=number of evaluable participants for each category.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 73
g/L
  Baseline for Week 12 (n=70) | 12.3 (1.4)
  Change at Week 12 (n=70) | 0.7 (1.2)
  Baseline for Week 24 (n=73) | 12.4 (1.5)
  Change at Week 24 (n=73) | 0.56 (1.1)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Regression Coefficient Between Change in Fatigue Score as Measured by the FACIT-F at Week 12 and 24 With Change in Disease Activity Parameters at Week 12 and 24
Description: Regression analysis between change in FACIT-F scale and change in following variable were assessed: DAS28-ESR (total score range: 0-9.4, higher score=more disease activity), Epworth sleepiness scale (total score range: 0-24, higher score=higher degree of sleepiness), back depression inventory (total score range: 0-63, score higher than 18 indicates moderate to severe symptoms of depression), serum hemoglobin, swollen joint count, morning stiffness (time taken to achieve maximum improvement), degree of pain (assessed on horizontal visual scale, 0=no pain; 10=maximum pain). The total score of the FACIT-F questionnaire ranges from 0=worse score to 52=better score. Regression coefficient (R) and coefficient of determination (R^2) were calculated. Difference (1-R^2)=the variation in the changes in fatigue not explained by independent variables, that is, independent contribution of these changes in fatigue to the assessment of RA. Only variables with available data were reported.
Time Frame: Week 12, 24
Population: Effectiveness analysis population. Here, N=number of participants analyzed for this measure.
Measure: Number; unit: unstandardized regression coefficient
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 84
unstandardized regression coefficient
  DAS-28 (Week 12) | -3.241
  DAS-28 (Week 24) | -2.596
  Serum hemoglobin (Week 12) | 0.335
  Serum hemoglobin (Week 24) | -0.242
  Swollen joint count (Week 12) | -0.333
  Swollen joint count (Week 24) | -0.600
  Morning stiffness (Week 12) | -0.559
  Morning stiffness (Week 24) | -0.718
  Degree of pain (Week 12) | -0.947
  Degree of pain (Week 24) | -0.839
  Sleepiness (Week 12) | -0.742
  Sleepiness (Week 24) | 1.193
  Depression (Week 12) | -0.714
  Depression (Week 24) | -0.777
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in DAS-28 at Week 12; Test type: Superiority or Other; p = 0.003, Regression, Linear
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in DAS-28 at Week 24; Test type: Superiority or Other; p = 0.006, Regression, Linear
Statistical Analysis 3: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in serum hemoglobin Week 12; Test type: Superiority or Other; p = 0.791, Regression, Linear
Statistical Analysis 4: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in serum hemoglobin Week 24; Test type: Superiority or Other; p = 0.847, Regression, Linear
Statistical Analysis 5: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in swollen joint count Week 12; Test type: Superiority or Other; p = 0.182, Regression, Linear
Statistical Analysis 6: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in swollen joint count Week 24; Test type: Superiority or Other; p = 0.022, Regression, Linear
Statistical Analysis 7: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in morning stiffness Week 12; Test type: Superiority or Other; p = 0.163, Regression, Linear
Statistical Analysis 8: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in morning stiffness Week 24; Test type: Superiority or Other; p = 0.115, Regression, Linear
Statistical Analysis 9: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in degree of pain Week 12; Test type: Superiority or Other; p = 0.037, Regression, Linear
Statistical Analysis 10: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in degree of pain Week 24; Test type: Superiority or Other; p = 0.044, Regression, Linear
Statistical Analysis 11: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in sleepiness at Week 12; Test type: Superiority or Other; p = 0.003, Regression, Linear
Statistical Analysis 12: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in sleepiness at Week 24; Test type: Superiority or Other; p = 0.001, Regression, Linear
Statistical Analysis 13: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 12 versus change in depression Week 12; Test type: Superiority or Other; p < 0.001, Regression, Linear
Statistical Analysis 14: Comparison: Rheumatoid Arthritis Participants; change in fatigue score at Week 24 versus change in depression at Week 24; Test type: Superiority or Other; p < 0.001, Regression, Linear

6. Secondary Outcome: Regression Coefficient Between Change in Hemoglobin Level at Week 12, 24 and Change in Disease Activity at Week 12 and 24
Description: Regression analysis between change in hemoglobin level and change in following variable were assessed: Epworth sleepiness scale (total score range: 0-24, higher score=higher degree of sleepiness), back depression inventory (total score range: 0-63, score higher than 18 indicates moderate to severe symptoms of depression), swollen joint count, morning stiffness (time taken to achieve maximum improvement), degree of pain (assessed on horizontal visual scale, 0=no pain; 10=maximum pain). Hemoglobin level was measure in g/L. The regression coefficient (R) and coefficient of determination (R^2) were calculated. Difference (1-R^2) indicates the variation in the changes in hemoglobin not explained by the independent variables, that is, independent contribution of these changes in hemoglobin to the assessment of RA. Only variables with available data were reported.
Time Frame: Week 12, 24
Population: Effectiveness analysis population. N=number of participants analyzed for this measure.
Measure: Number; unit: unstandardized regression coefficient
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 73
unstandardized regression coefficient
  Swollen joint count (Week 12) | -0.011
  Swollen joint count (Week 24) | 0.028
  Morning stiffness (Week 12) | 0.017
  Morning stiffness (Week 24) | -0.055
  Degree of pain (Week 12) | 0.021
  Degree of pain (Week 24) | 0.013
  Sleepiness (Week 12) | 0.004
  Sleepiness (Week 24) | 0.062
  Depression (Week 12) | -0.016
  Depression (Week 24) | -0.007
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in swollen joint count (Week 12); Test type: Superiority or Other; p = 0.678, Regression, Linear
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in swollen joint count (Week 24); Test type: Superiority or Other; p = 0.348, Regression, Linear
Statistical Analysis 3: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in morning stiffness (Week 12); Test type: Superiority or Other; p = 0.679, Regression, Linear
Statistical Analysis 4: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in morning stiffness (Week 24); Test type: Superiority or Other; p = 0.556, Regression, Linear
Statistical Analysis 5: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in degree of pain (Week 12); Test type: Superiority or Other; p = 0.692, Regression, Linear
Statistical Analysis 6: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in degree of pain (Week 24); Test type: Superiority or Other; p = 0.771, Regression, Linear
Statistical Analysis 7: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in sleepiness (Week 12); Test type: Superiority or Other; p = 0.878, Regression, Linear
Statistical Analysis 8: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in sleepiness (Week 24); Test type: Superiority or Other; p = 0.139, Regression, Linear
Statistical Analysis 9: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in depression score (Week 12); Test type: Superiority or Other; p = 0.249, Regression, Linear
Statistical Analysis 10: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in depression score (Week 24); Test type: Superiority or Other; p = 0.610, Regression, Linear

7. Secondary Outcome: Regression Coefficient Between Change in Hemoglobin Level at Week 12, 24 and Change in Disease Activity at Week 12 and 24 - Safety Population
Description: as for outcome 6
Time Frame: Week 12, 24
Population: Safety analysis population. Here, N=number of participants analyzed for this measure.
Measure: Number; unit: unstandardized regression coefficient
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 84
unstandardized regression coefficient
  Swollen joint count (Week 12) | 0.025
  Swollen joint count (Week 24) | 0.018
  Morning stiffness (Week 12) | 0.019
  Morning stiffness (Week 24) | -0.05
  Degree of pain (Week 12) | 0.022
  Degree of pain (Week 24) | 0.012
  Sleepiness (Week 12) | 0.002
  Sleepiness (Week 24) | 0.059
  Depression (Week 12) | -0.02
  Depression (Week 24) | -0.016
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in swollen joint count (Week 12); Test type: Superiority or Other; p = 0.257, Regression, Linear
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in haemoglobin levels versus change in swollen joint count (Week 24); Test type: Superiority or Other; p = 0.487, Regression, Linear
Statistical Analysis 3: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in morning stiffness (Week 12); Test type: Superiority or Other; p = 0.644, Regression, Linear
Statistical Analysis 4: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in morning stiffness (Week 24); Test type: Superiority or Other; p = 0.498, Regression, Linear
Statistical Analysis 5: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in degree of pain (Week 12); Test type: Superiority or Other; p = 0.650, Regression, Linear
Statistical Analysis 6: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in degree of pain (Week 24); Test type: Superiority or Other; p = 0.750, Regression, Cox
Statistical Analysis 7: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in sleepiness (Week 12); Test type: Superiority or Other; p = 0.936, Regression, Linear
Statistical Analysis 8: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in sleepiness (Week 24); Test type: Superiority or Other; p = 0.075, Regression, Linear
Statistical Analysis 9: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in depression score (Week 12); Test type: Superiority or Other; p = 0.098, Regression, Linear
Statistical Analysis 10: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in depression score (Week 24); Test type: Superiority or Other; p = 0.090, Regression, Linear

8. Secondary Outcome: Regression Coefficient Between Change in Hemoglobin Level at Week 12, 24 and Change in the Number of Swollen Joints (SJC 28) at Week 12 and 24 - Safety Population
Description: Regression analysis between the change in hemoglobin level and number of swollen joints was evaluated. Hemoglobin level was measure in g/L. The regression coefficient (R) and coefficient of determination (R^2) were calculated. Difference (1-R^2) indicates the variation in the changes in hemoglobin not explained by the independent variables, that is, independent contribution of these changes in hemoglobin to the assessment of RA. Only variables with available data were reported.
Time Frame: Week 12, 24
Population: Safety analysis population. N=participants who were evaluable for this outcome measure. n=number of participants evaluable in each category.
Measure: Number; unit: unstandardized regression coefficient
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 98
unstandardized regression coefficient
  Week 12 (n=91) | 0.186
  Week 24 (n=98) | 0.005
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in swollen joint count (Week 12); Test type: Superiority or Other; p = 0.077, Multiple Regression
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; change in hemoglobin levels versus change in swollen joint count (Week 24); Test type: Superiority or Other; p = 0.961, Multiple Regression

9. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count (SJC) at Week 12, 24
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, Week 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 83
swollen joints
  Baseline for Week 12 | 5.9 (4.6)
  Change at Week 12 | 1.9 (3.5)
  Baseline for Week 24 | 6.0 (4.6)
  Change at Week 24 | 1.8 (3.5)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count (SJC) at Week 12, 24 - Safety Population
Description: as for outcome 9
Time Frame: Baseline, Week 12, 24
Population: Safety population. N=participants who were evaluable for this outcome measure. n=number of participants evaluable in each category.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 113
swollen joints
  Baseline for Week 12 (n=109) | 5.7 (4.2)
  Change at Week 12 (n=109) | 2.1 (4.1)
  Baseline for Week 24 (n=113) | 5.9 (4.3)
  Change at Week 24 (n=113) | 1.8 (3.4)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 12, 24
Description: Duration of morning stiffness assessed as time taken to achieve maximum improvement from time participant rises. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 83
hours
  Baseline for Week 12 | 1.4 (2.7)
  Change at Week 12 | 0.5 (0.9)
  Baseline for Week 24 | 1.4 (2.8)
  Change at Week 24 | 0.4 (0.9)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 12, 24 - Safety Population
Description: as for outcome 11
Time Frame: Baseline, Week 12, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 112
hours
  Baseline for Week 12 (n=109) | 1.4 (2.5)
  Change at Week 12 (n=109) | 0.5 (0.8)
  Baseline for Week 24 (n=112) | 1.4 (2.5)
  Change at Week 24 (n=112) | 0.4 (0.8)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Pain Scores as Assessed by Visual Analogue Scale (VAS) at Week 12, 24
Description: Change from Baseline in 10 centimeter (cm) VAS pain score; 10-point pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Change = scores at observation minus score at Baseline. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 83
centimeter
  Baseline for Week 12 | 6.8 (2.1)
  Change at Week 12 | 2.57 (2.52)
  Baseline for Week 24 | 6.8 (2.1)
  Change at Week 24 | 2.57 (2.95)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Pain Scores as Assessed by Visual Analogue Scale (VAS) at Week 12, 24 - Safety Population
Description: Change from Baseline in 10 cm VAS pain score; 10-point pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Change = scores at observation minus score at Baseline. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 112
centimeter
  Baseline for Week 12 (n=107) | 6.9 (2.0)
  Change at Week 12 (n=107) | 2.59 (2.5)
  Baseline for Week 24 (n=112) | 6.9 (2.1)
  Change at Week 24 (n=112) | 2.69 (2.97)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Sleepiness Score as Assessed on Epworth Sleepiness Scale at Week 12, 24
Description: Degree of sleepiness was assessed by Epworth Sleepiness Scale. The Epworth Sleepiness Scale evaluates how likely a person is to doze off or fall asleep in 8 different sedentary situations, using for each item possible scores of 0 to 3 (0=never, 1=mild, 2=moderate and 3=severe). A final score is obtained between 0-24, where a higher score indicates a higher degree of sleepiness. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure. n=number of evaluable participants in each category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 83
score on a scale
  Baseline for Week 12 (n=82) | 6.0 (4.6)
  Change at Week 12 (n=82) | 5.4 (5.0)
  Baseline for Week 24 (n=83) | 6.1 (4.6)
  Change at Week 24 (n=83) | 5.3 (4.4)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p = 0.172, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.05, Regression, Logistic

16. Secondary Outcome: Change From Baseline in Sleepiness Score as Assessed on Epworth Sleepiness Scale at Week 12, 24 - Safety Population
Description: as for outcome 15
Time Frame: Baseline, Week 12, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 113
score on a scale
  Baseline for Week 12 (n=109) | 6.4 (5.0)
  Change at Week 12 (n=109) | 6.0 (4.4)
  Baseline for Week 24 (n=113) | 6.4 (4.5)
  Change at Week 24 (n=113) | 5.4 (4.5)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p = 0.162, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

17. Secondary Outcome: Change From Baseline in Depression Score as Assessed by the Beck Depression Inventory at Week 12, 24
Description: Mood assessed by the Beck Depression Inventory. The Beck Depression Inventory is a 21-item self-administered scale that evaluates severity of depression and is validated in Spanish on a 3 point scale (0=none to 3=severe). It measures the characteristic attitudes and symptoms of depression such as mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, etc. The total score ranges from 0 to 63. A score higher than 18 indicates moderate to severe symptoms of depression. Analysis include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis population. N=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 84
score on a scale
  Baseline for Week 12 | 17.4 (11.7)
  Change at Week 12 | 3.07 (9.09)
  Change at Week 24 | 3.5 (8.99)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.005, t-test, 2 sided

18. Secondary Outcome: Change From Baseline in Depression Score as Assessed by the Beck Depression Inventory at Week 12, 24 - Safety Population
Description: Mood assessed by the Beck Depression Inventory. The Beck Depression Inventory is a 21-item self-administered scale that evaluates severity of depression and is validated in Spanish on a 3 point scale (0=none to 3=severe). It measures the characteristic attitudes and symptoms of depression such as mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, etc. The total score ranges from 0 to 63. A score higher than 18 indicates moderate to severe symptoms of depression. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 113
score on a scale
  Baseline for Week 12 (n=111) | 18.3 (12.6)
  Change at Week 12 (n=111) | 3.5 (9.4)
  Baseline for Week 24 (n=113) | 18.5 (12.7)
  Change at Week 24 (n=113) | 3.89 (11.7)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.005, t-test, 2 sided

19. Secondary Outcome: Change From Baseline in Disease Activity Scale (DAS28) Score at Week 12, 24
Description: DAS28-4 erythrocyte sedimentation rate (ESR) was calculated from SJC and tender joint count (TJC) using 28 joints count, ESR millimeter per hour (mm/hr) and patient global assessment (PtGA) of disease activity (participant rated arthritis activity assessment). The DAS28-ESR score (14) was calculated using the following formula: DAS28 = 0.56 x (square root TJC) + 0.28 x (square root SJC) + 0.70 x [Ln(ESR)] + 0.014 x (PtGA).Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) less than or equal to (<=) 3.2 implied low disease activity and greater than (>)3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) less than (<)2.6 = remission. PtGA measured using a 100 mm VAS ranging from 0 = very good to 100 = very bad. Baseline data is reported separately for Weeks 12 and 24 to include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Effectiveness analysis: All participants who had at least one measurement of effectiveness subsequent to the start of tocilizumab (RoActemra) treatment were included. N=participants who were evaluable for this outcome measure. n=number of evaluable participants in each category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 71
score on a scale
  Baseline for Week 12 (n=66) | 3.0 (1.2)
  Change at Week 12 (n=66) | 2.53 (1.2)
  Baseline for Week 24 (n=71) | 2.7 (1.3)
  Change at Week 24 (n=71) | 2.73 (1.44)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 12 versus Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rheumatoid Arthritis Participants; Baseline for Week 24 versus Week 24; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

20. Secondary Outcome: Change From Baseline in Disease Activity Scale (DAS28) Score at Week 12, 24 - Safety Population
Description: DAS28-4 ESR was calculated from SJC and TJC using 28 joints count, ESR mm/hr and PtGA of disease activity (participant rated arthritis activity assessment). The DAS28-ESR score (14) was calculated using the following formula: DAS28 = 0.56 x (square root TJC) + 0.28 x (square root SJC) + 0.70 x [Ln(ESR)] + 0.014 x (PtGA).Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <=3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission. PtGA measured using a 100 mm VAS ranging from 0 = very good to 100 = very bad. Analysis include only those participants who had available data at Weeks 12 and 24, respectively.
Time Frame: Baseline, Week 12, 24
Population: Safety population. N=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 115
score on a scale
  Baseline for Week 12 | 5.6 (1.0)
  Change at Week 12 | 2.5 (1.1)
  Change at Week 24 | 2.7 (1.4)

21. Secondary Outcome: Percentage of Participants Achieving a Response According to European League Against Rheumatism (EULAR) Criteria at Week 12 and 24
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 reduction from Baseline. Participants with a score <=3.2 and reduction of >1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score <=5.1 with reduction of >0.6 to <=1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to <=1.2 points, or any score with reduction ≤0.6 points, were assessed as nonresponders with response recorded as 'none.' Participants with response is reported. DAS28 is described in outcome measure 19.
Time Frame: Week 12, 24
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 71
percentage of participants
  Good response at Week 12 (n=66) | 56.1
  Good response at Week 24 (n=71) | 62.0
  Moderate or good response at Week 12 (n=66) | 95.5
  Moderate or good response at Week 24 (n=71) | 93.0

22. Secondary Outcome: Percentage of Participants Achieving a Response According to European League Against Rheumatism (EULAR) Criteria at Week 12 and 24 - Safety Population
Description: as for outcome 21
Time Frame: Week 12, 24
Population: Safety population. N=participants who were evaluable for this outcome measure. n=number of evaluable participants in each category.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 115
percentage of participants
  Good response at Week 12 (n=85) | 51
  Good response at Week 24 (n=92) | 61
  Moderate or good response at Week 12 (n=85) | 95.3
  Moderate or good response at Week 24 (n=92) | 94.6

ADVERSE EVENTS:
Time Frame: Up to 1.5 year
Description: Safety analysis population: All participants who received at least one dose of the tocilizumab.
Groups:
- All Participants: Participants with moderate to severe RA who have been considered and proposed by the rheumatologist to start treatment with Tocilizumab (RoActemra) according to the indications of the summary of product characteristics of the product and the standard clinical practice of each participating center were followed-up for 6 months.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 3/120
Other Adverse Events (participants affected / at risk) | 27/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=120)
Arthritis infective (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Acute endocarditis (Infections and infestations) | 1
Pyelonephritis acute (Renal and urinary disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Rheumatoid lungs (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=120)
Aphthous stomatitis (Gastrointestinal disorders) | 7
Viral infection (Infections and infestations) | 6
Hypercholesterolemia (Metabolism and nutrition disorders) | 16
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.